CLINICAL TRIAL: NCT03550638
Title: The Efficacy and Safety Study on Endovascular Embolization of Intracranial Aneurysms With Coil System(Ton-bridgeMT)
Brief Title: Coil System(Ton-bridgeMT) for Endovascular Embolization of Cranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ2017001
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Coil system(Ton-bridgeMT)
  Interventions: Device: Coil system(Ton-bridgeMT)
- group B (Active Comparator): Axium Detachable Coil(Medtronic)
  Interventions: Device: Axium Detachable Coil(Medtronic)

INTERVENTIONS:
Device: Coil system(Ton-bridgeMT) — 1. It consists of a push system with a development mark, and a Detachable platinum-tungsten alloy coil which is connected to the push system. It can be used for embolization of intracranial aneurysms, and other neurovascular abnormalities, such as arteriovenous malformation and arteriovenous fistula.
  Arms: group A
Device: Axium Detachable Coil(Medtronic) — 2. It is made up of a push system with a development mark, a platinum-tungsten alloy embolized coil connected to the push system and a manual release device for releasing the coil from the distal end of the push system. It is mainly used for embolization of intracranial aneurysms, and other neurovascular abnormalities, such as arteriovenous malformation and arteriovenous fistula.
  Arms: group B

SUMMARY:
The study is a prospective, multi-center, randomized, open, parallel positive control, non-inferiority trial. Patients are randomized 1:1 to either Coil System(Ton-bridgeMT) or Axium Detachable Coil(Medtronic).

The purpose of this study is to assess the safety and effectiveness of the Coil System(Ton-bridgeMT) in the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Subject has a target intracranial aneurysm (IA) diagnosed by DSA, and intended to be embolised with coil system.
* Subject or guardian is able to understand the purpose of study, agrees to comply with protocol requirements and has provided written informed consent.

Exclusion Criteria:

* Subject is diagnosed as multiple aneurysms.
* Subject is diagnosed as intracranial bulloid, fusiform, false, dissectimng, infective aneurysm or with arteriovenous malformation.
* mRS score≥3.
* Hunt and Hess classification≥4.
* Subject has emergency ruptured aneurysms and needs assisting stent.
* The target aneurysm has received endovascular embolization or surgical treatment.
* The aneurysm carrier artery has severe stenosis.
* PLT<60×109/L or INR>1.5.
* Subject has nonfunction of important organs or other severe diseases.
* Major surgery in the last 30 days, or intending to receive surgical treatment in 90 days after enrollment.
* Subject is allergic to antiplatelet drugs, anticoagulants, anesthetics, contrast agents or any related contraindication.
* History of allergies to platinum and tungsten.
* Expected life <12 months.
* Pregnant or lactating women.
* Subject has participated in any other drug or medical device clinical trials in 1 month before writting informed consent .
* Other circumstances judged by researchers are not suitable for enrollment .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
success rate of occlusion | 180 day
  Number of aneurysms(Raymond Ⅰ and Ⅱ)/number of overall aneurysms*100%

SECONDARY OUTCOMES:
success rate of occlusion | intraoperation
  Number of aneurysms(Raymond Ⅰ and Ⅱ)/number of overall aneurysms*100%
Recurrence rate | 180 day
  2. Number of patients with recurrent aneurysms/ number of overall patients*100%

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital of Shangha
Locations (12):
- China (12):
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Jiangsu Province Hospital, Nanjin, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, Xi’an, Shanxi
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hanzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No